CLINICAL TRIAL: NCT01650922
Title: Molecular Genetic Studies of Childhood Brain Tumors and Blood Samples
Status: Completed | Type: Observational
Sponsor: Stanford University (Other)
Responsible Party: Sponsor
Other Study IDs: PEDSBRN0004; 96447; PEDSBRN0004
Record Dates: First submitted 2012-07-24; First posted 2012-07-26 (Estimated); Last update posted 2012-07-26 (Estimated); Status verified 2012-07

CONDITIONS: Brain Cancer
MeSH Terms: conditions — Brain Neoplasms | interventions — Phlebotomy; Biopsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — the investigators will sample a single blood sample or buccal swab and if obtained at the time of diagnosis, brain tumor biopsy.

INTERVENTIONS:
Procedure: phlebotomy
Procedure: biopsy

SUMMARY:
To look for patterns of polymorphisms in DNA repair in both germline and tumor cells samples.

ELIGIBILITY:
Inclusion Criteria:Pediatric cancer patients diagnosed with brain tumors

Max Age: 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Pediatric cancer patients diagnosed with brain tumors
Sampling Method: Non-Probability Sample
Enrollment: 4 (Actual)
Dates: Start 2005-09; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James M Ford, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States